CLINICAL TRIAL: NCT02020993
Title: The Prognostic Value of Urine NT-ProBNP in Neonatal Respiratory Distress
Brief Title: Urine NT-ProBNP in Neonatal Respiratory Distress
Acronym: NT-proBNP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Duran Yildiz, MD, Ankara University
Other Study IDs: NT-proBNP Trial
Record Dates: First submitted 2013-12-03; First posted 2013-12-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Neonatal Respiratory Distress
Keywords: Nt-proBNP, newborn, preterm
MeSH Terms: conditions — Pulmonary Atelectasis; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine NT-proBNP
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Respiratory distress group: Newborns with respiratory distress will constitute the study group. All patients will be evaluated by Urine NT-proBNP and echocardiography on postnatal days 1-2 and 5-7.
- Control Group: Newborns without any respiratory and cardiac diseases will constitute the control group, and will be evaluated by urine Nt-proBNP and echocardiography on postnatal days 1-2 and 5-7.

SUMMARY:
There is a need for a biochemical marker in addition to clinical condition which will help the physician to understand the clinical progress of the disease.

Urine Nt-proBNP, which does not need any blood sampling and can be collected easily, has not been evaluated for respiratory distress in newborn.

The investigators aim to evaluate the prognostic value of urine NT-proBNP in respiratory diseases in newborns by a controlled trial.

DETAILED DESCRIPTION:
Neonatal diseases such as respiratory distress and transient tachypnea of newborn may require high level of intensive care. On the other hand, some minor difficulties in respiration can resolve within hours. Therefore, there is a need for a biochemical marker in addition to clinical condition which will help the physician to understand the clinical progress of the disease.

Serum NT-ProBNP level has been evaluated in transient tachypnea of newborn and found compatible with the clinical progress. Urine NT-proBNP has recently been evaluated in patent ductus arterioses and found compatible with the cardiac progress. However, urine Nt-proBNP, which does not need any blood sampling and can be collected easily, has not been evaluated for respiratory distress in newborn.

The investigators aim to evaluate the prognostic value of urine NT-proBNP in respiratory diseases in newborns by a controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* study group; newborns who are admitted to the neonatal intensive care unit within first 2 days of life and have transient tachypnea of newborn or respiratory distress syndrome signed informed consent form
* Control Group: Newborns without any respiratory distress

Exclusion Criteria:

* any cardiac anomaly sepsis acute renal insufficiency syndromic cases low APGAR score at 5th minute (<7) lung malformations no informed consent inability in collection of urine

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Newborns with first postnatal 2 days with or without respiratory distress
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
severity of respiratory distress | 7 days
  Severity of respiratory distress will be evaluated by requirement of supportive treatment such as continuous positive airway pressure, need of intubation, mechanical ventilation and duration of support (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Begüm Atasay, Professor, Principal Investigator — Ankara University
Locations (1):
- Ankara University, Ankara, Ankara, Turkey (Türkiye)